CLINICAL TRIAL: NCT03472456
Title: Articaine or Eugenol: a Study on the Choice of Endodontic Medication in the Emergency Management of Irreversible Pulpitis of a Mature Permanent Tooth
Brief Title: Endodontic Medications for Irreversible Pulpitis: Articaine or Eugenol?
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6953
Record Dates: First submitted 2018-02-12; First posted 2018-03-21 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Pulpitides; Endodontic Inflammation; Toothaches; Operative Dentistry
MeSH Terms: conditions — Pulpitis; Toothache | interventions — Compliance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Articaïne
  Interventions: Drug: Implementation of a pulp medication in compliance with the dental emergency management protocol: articaïne
- Eugénol
  Interventions: Drug: Implementation of a pulp medication in compliance with the dental emergency management protocol: eugenol

INTERVENTIONS:
Drug: Implementation of a pulp medication in compliance with the dental emergency management protocol: articaïne — Implementation of a pulp medication in compliance with the dental emergency management protocol: articaïne
  Groups: Articaïne
Drug: Implementation of a pulp medication in compliance with the dental emergency management protocol: eugenol — Implementation of a pulp medication in compliance with the dental emergency management protocol: eugenol
  Groups: Eugénol

SUMMARY:
The objective of the study is to determine which of the two commonly used endodontic medications (Eugenol VS Articaine) is most effective in controlling postoperative pain in irreversible pulpitis of the mature permanent tooth in adults. To do so, an assessment of the pain felt by patients will be carried out a few days apart. The supposed results are that the medications are equivalent in terms of effectiveness on the pain, but could then present different economic arguments

DETAILED DESCRIPTION:
In irreversible pulpitis of the mature permanent tooth, the enrolled patients receive endodontic medications (Eugenol or Articaine) in order to determine which one is the more efficient to control the pain.

These patients would have received the same medication without this study. That's why this is an obsevationnal study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, major, affiliated to a social health insurance scheme
* Patient having agreed to participate in the study
* Urgent consultant patient for irreversible pulpitis
* Patient understanding French

Exclusion Criteria:

* Refusal of the patient to participate in the study
* Impossibility of performing the surgical procedure
* Impossibility to give the subject information enlightened (difficulty of understanding ...)
* Subject under the protection of justice, or under guardianship
* General contraindication to endodontic treatment in 2 sessions (high risk of infectious endocarditis, for example)
* Chronic intake of analgesic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the University Hospital (Dental Service) of Strasbourg (HUS)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2018-03-22 (Actual); Study Completion 2019-10-24 (Actual)

PRIMARY OUTCOMES:
Pain evolution (decrease or increase the intensity of the pain) | 7 days
  Evolution of pain (using a score of 0 to 10)

CONTACTS AND LOCATIONS:
Overall Officials: Damien OFFNER, Principal Investigator — Les Hôpitaux Universitaires de Strasbourg
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided